CLINICAL TRIAL: NCT03967626
Title: Practical Efficiency of Coupling Targeted Temperature Management to Brain Temperature Rather Than Systemic Temperature in Severe Brain Injury (BRAIN TTM)
Brief Title: Efficiency of Coupling Targeted Temperature Management to Brain Temperature in Severe Brain Injury
Acronym: BRAINTTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NED_2019_7
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2024-06

CONDITIONS: Brain Injuries
Keywords: Temperature targeted management (TTM); close loop; brain temperature; cerebral temperature; systemic temperature; neuroprotection; fever control
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: * experimental group: CCT (cerebral temperature target) performed by the external cooling device on the TC measured by the PIC/TC sensor (PIC:intracranial pressure)
  * control group: CCT performed by the external cooling device on the TS, measured by a bladder sensor (coupled to the vesal probe, according to the standard service protocol).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerebral temperature target (Experimental): CCT performed by the external cooling device with cerebral temperature target, measured by a intracranial sensor (coupled to the intracranial pressure device)
  Interventions: Device: external cooling with the xxxxx device
- Systemic temperature target (Active Comparator): CCT performed by the external cooling device with systemic temperature target, measured by a bladder sensor (coupled to the vesal probe, according to the standard service protocol).
  Interventions: Device: external cooling with the xxxxx device

INTERVENTIONS:
Device: external cooling with the xxxxx device — external cooling with the xxxxx device

SUMMARY:
In severe brain-injured patients, it is recommended to strictly control the fever in order to limit brain damage (objective of neuroprotection) via the targeted temperature management (TTM). In the guidelines, the target temperature is the systemic temperature, just for practical reasons (brain temperature not being monitored in most polyvalent ICU). However, in NICU, the brain temperature is monitored routinely via the Intra-Cerebral Pressure (ICP) sensor. Since in the febrile brain-injured patients the objective of the TTM is neuroprotection, it would be more appropriate to target temperature control over the cerebral temperature.

The objective of this study is to evaluate the efficacy of TTM directly coupled to the brain temperature.

Adult patients with brain injury requiring ICP monitoring (Pressio 2, Sophysa France) and fever requiring TTM (cerebral greater than or equal to 38.5 °C) will be enrolled. The TTM will be carried out according to the usual methods of the investigator's service: external cooling devices coupled with cerebral temperature (Artic Sun, Bard France), including two phases: the cooling phase (H0 to H3) and the maintenance phase (from H3 to the end of the cooling).

Two groups will be formed. In the interventional group, coupling of the TTM will be carried out to the cerebral temperature. In the control group, coupling of the TTM will be carried out to the systemic temperature measured at the bladder site.

The primary outcome will be the percentage of time during which the cerebral temperature will be measured within recommended target temperature range (i.e. 36 to 37 °C) during the maintenance phase (H3 to H12): comparison of averages. Cerebral hemodynamic parameters (ICP, transcranial doppler, and brain tissue oxygen partial pressure if available) will also be collected, in order to be correlated with the delta temperature (cerebral temperature minor systemic temperature).

No medical device will be put in place specifically for the need of the study.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years of age or older
* hospitalized patient in neuro-resuscitation with peak monitoring with cerebral temperature measurement by an intra-parenchymal sensor (Sophysa®)
* patient in hyperthermia (TC ≥ 38.5 °c) and in a situation of brain pain

Exclusion Criteria:

* patient benefiting from a legal protection measure
* pregnant or breastfeeding woman
* previous participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
The percentage of time with brain temperature between (36.5 ± 0.5 °C) | 12 hours
  The percentage of time during which the measured brain temperature is included in the target temperature range (36.5 ± 0.5 °C), during the maintenance phase (averages comparison).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation Adolphe Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stephan S, Cohen F, Salviat F, Thevenin S, Devys JM, Cochereau I, Gabison E. Evaluation of the impact of intensive care support for COVID-19 on the ocular surface in a prospective cohort of 40 eyes. Ocul Surf. 2021 Oct;22:13-14. doi: 10.1016/j.jtos.2021.06.008. Epub 2021 Jun 23. No abstract available. PMID 34174393